CLINICAL TRIAL: NCT06950073
Title: CUratively Intended Thoracic REirradiation: An Observational Study of High-dose Reirradiation of Thoracic Tumours: A Multicentre Prospective Registration Protocol
Brief Title: Curatively Intended Thoracic Reirradiation
Acronym: CureLung
Status: Not yet recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: Curelung2025; R374-A22286 (Other Grant/Funding Number: Danish Cancer Society)
Record Dates: First submitted 2025-04-14; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-03

CONDITIONS: Radiotherapy Side Effect; Radiation Toxicity; Oncology; Lung Cancer; Thoracic Cancer
Keywords: Reirradiation
MeSH Terms: conditions — Radiation Injuries; Neoplasms; Lung Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with thoracic cancer elegible for reirradation.: Recurrent lung cancer, new primary lung cancer, solitary lung metastasis
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Radiotherapy is offered in the same dose to all patients eligible to reirradiation no matter if they are enrolled in the study or not. Meaning no intervention is done. This is a registration study.

SUMMARY:
The number of long-term lung cancer (LC) survivors increases, however many patients are diagnosed with recurrent or new thoracic cancers. High-dose reirradiation (reRT) is promising but associated with high severe toxicity rates. Existing studies are small lacking high-quality data, with no clear correlation between toxicity risk and delivered radiotherapy (RT) dose.

This Danish multicentre prospective cohort study aims to provide a framework for collecting radiotherapy-related toxicity data, loco-regional control, and overall survival data for patients with thoracic cancer undergoing reirradiation; with the ultimate aim of providing safe reirradiation to more patients.

As a secondary aim, guidelines for dose accumulation and provisional constraints for the organs at risk will be used to establish a uniform treatment strategy for reirradiation.

The CURE Lung trial will provide high-impact, globally missing data. This project will ensure full utilization of and learning from the trial, adding SDM, PROMs, and modality referral to the trial. It will model the correlation between toxicity burden and doses, enabling individualized reRT with optimized dose prescription based on toxicity risk and patient preferences, and assisting in the decision-making on the prescription dose and optimal modality. This will ensure safe reRT for the increasing number of long-term LC survivors.

DETAILED DESCRIPTION:
1. BACKGROUND:

   The number of long-term survivors is increasing for thoracic cancers, however, a significant proportion of lung cancer (LC) patients treated with curatively intended radiotherapy (RT) may experience locoregional recurrence or develop a new cancer. This highlights the need for effective local treatment options. Repeated high-dose RT (reRT) is a promising approach gaining traction in clinical practice. At Aarhus University Hospital (AUH), the fraction of LC patients offered curative reRT has increased from 4% in 2015 to 13% in 2024. The overall survival (OS) of reirradiated recurrent or new LC range from 7-14 months (from time of reirradiation) and depends on a variety of parameters, including tumour dose and PTV volume. ReRT has been linked to high rates of severe toxicity, leading to some patients not being offered curative reRT. Establishing solid evidence of the risks associated with reRT is crucial to offering these patients reRT on an equal footing with patients treated for their first cancer. Former studies on reRT of LC include a median of 40 (maximum 102) patients16, with diverse results on OS and no clear correlations between toxicity risk and cumulative (summed) RT doses.
2. AIM:

   Establish a framework for LC reRT based on data from CURE Lung to support clinical and shared decision-making (SDM). Four sub-studies obtain this:

   2.1 Establish a national infrastructure for reRT and implement decision-making tools to guide patient referrals to specialised modalities like proton therapy and MR-linac, ensuring optimal treatment modality selection to reRT for the individual patient.

   2.2 Integrate and analyse Patient Reported Outcome Measures (PROM), Quality of Life (QoL), and decision regret data in CURE Lung. Mapping of the patient's self-reported symptoms and correlation to toxicity data ensures an optimal overview of total disease burden and informs which patients are candidates for reRT.

   2.3 Establish and evaluate SDM focusing on the clinical risk assessment and the patient's wishes as tools for optimal patient involvement. SDM will improve the participants' knowledge, and accuracy of risk perceptions, and help them choose the best treatment, minimizing regret and improving QoL.

   2.4 Build models correlating patient- and physician-reported toxicity to RT doses, considering prior treatments, co-morbidity, and QoL to inform decision-making. This will provide dose limits for reRT, allowing individualised dose prescriptions based on toxicity risk, comorbidities and prior treatments.
3. HYPOTHESES:

   Primary hypothesis:

   - Cumulative radiation dose is related to radiotherapy-related toxicity for patients undergoing thoracic reirradiation

   Secondary hypothesis:

   - Curative reirradiation is feasible and safe for a selected patient cohort when delivered based on strict dose limits
4. PATIENTS:

   Recurrent or new LC, or solitary oligo lung metastases. The investigators plan for 500 patients in 3-4 years. Annually, approximately 100-150 patients are expected from the seven Danish RT centres based on a recent comprehensive national audit of RT retreatment numbers and sites.
5. TRIAL DESIGN AND DATA COLLECTION:

   This is a multicentre prospective registration protocol.

   The trial is based on a high mandatory standard being mandatory for participation with 1) 3D dose summation, 2) data on previous RT, systemic treatments, surgery, comorbidity and G3-4 thoracic toxicity collected at baseline, 3) prospective clinical follow-up with G2-5 toxicity scoring, and thoracic CT-imaging, performed every three months until two years and bi-annually until five years enabling reliable longitudinal toxicity scoring, and 4) pre-trial QA consisting of image registration, treatment planning and healthy tissue delineation.

   Toxicity and patient-reported outcomes (PROM) will be monitored during and up to 5 years after treatment using common terminology criteria for adverse events (CTCAE) and the European Organisation for Research and Treatment of Cancer (EORTC) QoL questionnaires (QLQ-C30 and LC13). Central databases will be used for clinical (Redcap) and dosimetric (dcmcollab) data collection.
6. PERSPECTIVES:

The CURE Lung trial will yield internationally high-impact results. The trial is based on state-of-the-art treatment delivery, dose accumulation, and clinical data collection, ensuring exceptional data quality for modelling studies. The trial data will be unique in patient numbers and data quality. Similar data are not available Worldwide. The current project will ensure full utilisation of and learning from the trial, adding SDM, PROMs, referral to specialised modalities, and high-level QA to the trial. It will enable modelling the correlation between toxicity burden and individual patient doses, paving the way for individualised reRT with optimised dose prescription based on toxicity risk and patient preferences, and assisting in the decision-making on the prescription dose and optimal modality. This will ensure safe reRT for the increasing number of long-term LC survivors.

Results will be published in scientific international journals (Radiother Oncol, Int J Radiat Oncol Biol Phys, J Clin Oncol, and J Thorac Oncol), and presented at international conferences and Danske Kræftforskningsdage.

The findings may apply to reRT for other cancers, benefitting all Danish patients. The project underpins the new work package for reRT under the Danish Comprehensive Cancer Center for RT (DCCC-RT), aiming to collect and standardize national reRT data.

ELIGIBILITY:
Inclusion Criteria:

* Radiotherapy of thoracic lesion(s) (loco-regional lung cancer recurrence, new primary lung cancer, or solitary oligo metastasis) with the aim of long-term local control.
* Reirradiation type 1 or type 2, i.e. previous radiotherapy to the thorax as per ESTRO-EORTC consensus definition of reirradiation [Andratschke 2022]. For the sake of this study, multiple treatments to the lungs will be classified as type 2 reirradiation.
* Verification of malignancy based on biopsy. If no biopsy is available, the decision of reirradiation should be agreed upon in a multidisciplinary conference.
* Available digital dose plan(s) from former radiotherapy course(s) (DICOM files) - note that multiple re-treatments are allowed.
* Adequate lung function to tolerate treatment, at the discretion of the treating physician.
* Ability to complete a radiotherapy course with the aim of local control.
* ECOG Performance status 0-2.
* Estimated life expectancy ≥ 6 months
* Age ≥18 years
* Signed informed consent

Exclusion Criteria:

* Uncontrolled other malignancy.
* The primary and the reirradiation treatment may not be quasi-simultaneous (i.e. the two treatments should be planned independently)
* Pregnancy
* Radiotherapy to a minimum CTV mean dose of 45 Gy for SCLC and 50 Gy for NSCLC and oligometastatic lesions. Treatment schedule according to local protocols and treating physician preference.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Recurrent or new LC, or solitary oligo lung metastases. We plan for 500 patients in 3-4 years. Annually, approximately 100-150 patients are expected from the seven Danish RT centres based on a recent comprehensive national audit of RT retreatment numbers and sites.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2035-05-01 (Estimated); Study Completion 2035-05-01 (Estimated)

PRIMARY OUTCOMES:
Toxicity grade 4-5 | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Radiotherapy-related toxicity using the Common Terminology Criteria for Adverse Events (CTCAE) grade 4 - 5 one year after start of radiotherapy

SECONDARY OUTCOMES:
Overall survival | From date of enrollment until the date of documented death
  The length of time from the start of radiotherapy, that patients are still alive.
Freedom from progressive disease | From date of enrollment until the date of documented progression
  The length of time from the start of radiotherapy, that a patient lives with the disease without it getting worse
Patterns of failure | From date of enrollment until the date of documented recurrence
  If recurrence is diagnosed, where have the disease reappeared?
Acute radiotherapy-related toxicity grade 2 - 5 | Up to 6 months from the start of reirradiation
  Using the Common Terminology Criteria for Adverse Events (CTCAE) toxicity grade 2 - 5
Late radiotherapy-related toxicity grade 3 - 5 | From 6 months after the start of reirradiation and through study completion, assessed up to 60 months
  Using the Common Terminology Criteria for Adverse Events (CTCAE) toxicity grade 3-5
Radiotherapy treatment compliance | Through study completion, assessed up to 60 months
  The extent to which a person's behavior follows medical advice or corresponds with recommendations from the health care provider.
Quality of Life (QoL) | Baseline, at 3 months, and each year through study completion
  The European Organisation for Research and Treatment of Cancer (EORTC) QoL questionnaires C30 (general module) and LC13 (lung cancer-specific module) will be used to evaluate QoL and symptoms.
Patient reported outcome measures (PROM) | Baseline, at 3 months, and each year through study completion
  The EuroQol 5-level EQ-5D version (EQ-5D-5L) questionnaire will be used to describe the health state of the patients.
Decision regret according to the Ottawa Hospital scale | Baseline, at 3 months, and each year through study completion
  Decision regret is a negative emotion involving distress or remorse following a decision related to the treatment

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Abusaris H, Storchi PR, Brandwijk RP, Nuyttens JJ. Second re-irradiation: efficacy, dose and toxicity in patients who received three courses of radiotherapy with overlapping fields. Radiother Oncol. 2011 May;99(2):235-9. doi: 10.1016/j.radonc.2011.03.010. Epub 2011 Apr 15. PMID 21497928
- [Background] Amini A, Yang J, Williamson R, McBurney ML, Erasmus J Jr, Allen PK, Karhade M, Komaki R, Liao Z, Gomez D, Cox J, Dong L, Welsh J. Dose constraints to prevent radiation-induced brachial plexopathy in patients treated for lung cancer. Int J Radiat Oncol Biol Phys. 2012 Mar 1;82(3):e391-8. doi: 10.1016/j.ijrobp.2011.06.1961. PMID 22284035
- [Background] Andratschke N, Willmann J, Appelt AL, Alyamani N, Balermpas P, Baumert BG, Hurkmans C, Hoyer M, Langendijk JA, Kaidar-Person O, van der Linden Y, Meattini I, Niyazi M, Reynaert N, De Ruysscher D, Tanadini-Lang S, Hoskin P, Poortmans P, Nieder C. European Society for Radiotherapy and Oncology and European Organisation for Research and Treatment of Cancer consensus on re-irradiation: definition, reporting, and clinical decision making. Lancet Oncol. 2022 Oct;23(10):e469-e478. doi: 10.1016/S1470-2045(22)00447-8. PMID 36174633
- [Background] Ang KK, Price RE, Stephens LC, Jiang GL, Feng Y, Schultheiss TE, Peters LJ. The tolerance of primate spinal cord to re-irradiation. Int J Radiat Oncol Biol Phys. 1993 Feb 15;25(3):459-64. doi: 10.1016/0360-3016(93)90067-6. PMID 8436524
- [Background] Ang KK, Jiang GL, Feng Y, Stephens LC, Tucker SL, Price RE. Extent and kinetics of recovery of occult spinal cord injury. Int J Radiat Oncol Biol Phys. 2001 Jul 15;50(4):1013-20. doi: 10.1016/s0360-3016(01)01599-1. PMID 11429229
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Yokoi T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Wadsworth C, Melillo G, Jiang H, Huang Y, Dennis PA, Ozguroglu M; PACIFIC Investigators. Durvalumab after Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Nov 16;377(20):1919-1929. doi: 10.1056/NEJMoa1709937. Epub 2017 Sep 8. PMID 28885881
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Kurata T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Faivre-Finn C, Reck M, Vansteenkiste J, Spigel DR, Wadsworth C, Melillo G, Taboada M, Dennis PA, Ozguroglu M; PACIFIC Investigators. Overall Survival with Durvalumab after Chemoradiotherapy in Stage III NSCLC. N Engl J Med. 2018 Dec 13;379(24):2342-2350. doi: 10.1056/NEJMoa1809697. Epub 2018 Sep 25. PMID 30280658
- [Background] Auperin A, Le Pechoux C, Rolland E, Curran WJ, Furuse K, Fournel P, Belderbos J, Clamon G, Ulutin HC, Paulus R, Yamanaka T, Bozonnat MC, Uitterhoeve A, Wang X, Stewart L, Arriagada R, Burdett S, Pignon JP. Meta-analysis of concomitant versus sequential radiochemotherapy in locally advanced non-small-cell lung cancer. J Clin Oncol. 2010 May 1;28(13):2181-90. doi: 10.1200/JCO.2009.26.2543. Epub 2010 Mar 29. PMID 20351327
- [Background] Badiyan SN, Rutenberg MS, Hoppe BS, Mohindra P, Larson G, Hartsell WF, Tsai H, Zeng J, Rengan R, Glass E, Katz S, Vargas C, Feigenberg SJ, Simone CB 2nd. Clinical Outcomes of Patients With Recurrent Lung Cancer Reirradiated With Proton Therapy on the Proton Collaborative Group and University of Florida Proton Therapy Institute Prospective Registry Studies. Pract Radiat Oncol. 2019 Jul-Aug;9(4):280-288. doi: 10.1016/j.prro.2019.02.008. Epub 2019 Feb 23. PMID 30802618
- [Background] Basch E, Iasonos A, McDonough T, Barz A, Culkin A, Kris MG, Scher HI, Schrag D. Patient versus clinician symptom reporting using the National Cancer Institute Common Terminology Criteria for Adverse Events: results of a questionnaire-based study. Lancet Oncol. 2006 Nov;7(11):903-9. doi: 10.1016/S1470-2045(06)70910-X. PMID 17081915
- [Background] Basch E. The missing voice of patients in drug-safety reporting. N Engl J Med. 2010 Mar 11;362(10):865-9. doi: 10.1056/NEJMp0911494. No abstract available. PMID 20220181
- [Background] Becerra Perez MM, Menear M, Brehaut JC, Legare F. Extent and Predictors of Decision Regret about Health Care Decisions: A Systematic Review. Med Decis Making. 2016 Aug;36(6):777-90. doi: 10.1177/0272989X16636113. Epub 2016 Mar 14. PMID 26975351
- [Background] Bellera CA, Rainfray M, Mathoulin-Pelissier S, Mertens C, Delva F, Fonck M, Soubeyran PL. Screening older cancer patients: first evaluation of the G-8 geriatric screening tool. Ann Oncol. 2012 Aug;23(8):2166-2172. doi: 10.1093/annonc/mdr587. Epub 2012 Jan 16. PMID 22250183
- [Background] Bergman B, Aaronson NK, Ahmedzai S, Kaasa S, Sullivan M. The EORTC QLQ-LC13: a modular supplement to the EORTC Core Quality of Life Questionnaire (QLQ-C30) for use in lung cancer clinical trials. EORTC Study Group on Quality of Life. Eur J Cancer. 1994;30A(5):635-42. doi: 10.1016/0959-8049(94)90535-5. PMID 8080679
- [Background] Bertelsen AS, Schytte T, Moller PK, Mahmood F, Riis HL, Gottlieb KL, Agergaard SN, Dysager L, Hansen O, Gornitzka J, Veldhuizen E, ODwyer DB, Christiansen RL, Nielsen M, Jensen HR, Brink C, Bernchou U. First clinical experiences with a high field 1.5 T MR linac. Acta Oncol. 2019 Oct;58(10):1352-1357. doi: 10.1080/0284186X.2019.1627417. Epub 2019 Jun 26. PMID 31241387
- [Background] Binkley MS, Hiniker SM, Chaudhuri A, Maxim PG, Diehn M, Loo BW Jr, Shultz DB. Dosimetric Factors and Toxicity in Highly Conformal Thoracic Reirradiation. Int J Radiat Oncol Biol Phys. 2016 Mar 15;94(4):808-15. doi: 10.1016/j.ijrobp.2015.12.007. Epub 2015 Dec 17. PMID 26831903
- [Background] Bjordal K, de Graeff A, Fayers PM, Hammerlid E, van Pottelsberghe C, Curran D, Ahlner-Elmqvist M, Maher EJ, Meyza JW, Bredart A, Soderholm AL, Arraras JJ, Feine JS, Abendstein H, Morton RP, Pignon T, Huguenin P, Bottomly A, Kaasa S. A 12 country field study of the EORTC QLQ-C30 (version 3.0) and the head and neck cancer specific module (EORTC QLQ-H&N35) in head and neck patients. EORTC Quality of Life Group. Eur J Cancer. 2000 Sep;36(14):1796-807. doi: 10.1016/s0959-8049(00)00186-6. PMID 10974628